CLINICAL TRIAL: NCT02609022
Title: A First-in-human and Proof-of-concept Study to Assess the Safety, Tolerability and Immunogenic Response of CV-MG01, Acetylcholine Receptor Mimetic Peptides, as Potential Therapeutic Vaccine, in Patients With Myasthenia Gravis
Brief Title: Safety, Tolerability and Immunogenic Response of CV-MG01 in Patients With Myasthenia Gravis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CuraVac (Industry)
Collaborators: Aepodia (Industry); University Hospital, Antwerp (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV-0002; 2015-002880-41 (EudraCT Number)
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; CV-MG01 therapeutic vaccine; Acetylcholine receptor mimetic peptides; Safety; Immunogenic response; First-in-Human; Proof-of-Concept; Myasterix
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CV-MG01 (Experimental): The therapeutic vaccine candidate, CV-MG01 comprises two short synthetic peptides separately conjugated to a carrier protein for the potential treatment of myasthenia gravis
  Interventions: Biological: CV-MG01
- Placebo (Placebo Comparator): Aluminium hydroxide adjuvant alone
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CV-MG01 — 3 consecutive subcutaneous injections of CV-MG01. The three injections are planned for each patient on Days 1, 29 (+/- 3 days) and 85 (+/- 7 days), respectively.
  Two dose levels: low and high dose.
  Arms: CV-MG01
Biological: Placebo — 3 consecutive subcutaneous injections of placebo. The three injections are planned for each patient on Days 1, 29 (+/- 3 days) and 85 (+/- 7 days), respectively.
  Arms: Placebo

SUMMARY:
Study CV-0002 is the first clinical trial administering CV-MG01 in humans. This clinical trial is a safety and proof-of-concept study (proof of mechanism of action) intended to assess the safety, tolerability and immunogenic response following 3 subcutaneous injections of CV-MG01 as a potential therapeutic vaccine / active immunotherapy in myasthenia gravis (MG) patients.

DETAILED DESCRIPTION:
Part A of the trial has been designed as a human safety pharmacology and therapeutic exploratory, parallel group, randomised, placebo-controlled, single centre, Investigator and subject-blind study using adaptive dose and sample size approaches.

At the end of part A of the present study, all patients, including those receiving placebo, will be monitored in an open label, long-term safety follow-up part B of the study to assess the treatment effects over time.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, with ocular and generalised myasthenia gravis (grade 1-2-3).
* Between the ages of 18 and 64 years, inclusive, at the time of the first injection.
* A Body Mass Index (BMI) between 18 and 35 kg/m2, inclusive.
* Patient with positive antibodies to AChR based on radioimmunoassay(RIA) (AChRAb ≥ 1 nmol/l); if available, historical data on AChR Ab levels over the last 2 years will be collected in the study records.
* Patient may use corticosteroid treatment, equivalent to a daily dose of 30 mg prednisone or lower and stable (dose +/- 5 mg) during the 3 months before participation.
* Patient may use one immunosuppressive drug with or without concomitant use of corticosteroid, providing that the dosage has been stable/unchanged for 3 months before participation.
* Blood pressure and heart rate (supine & standing) within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by the relevant Ethics Committee (EC) governing the site.

Exclusion Criteria:

* MG patients of Grade 4 or 5 based on myasthenia gravis foundation of America (MGFA) classification.
* Patients with history or presence of a primary or recurrent malignant disease including the presence or history of a thymoma.
* Thymectomy planned during part A of the study period or performed within 1 year prior to the first dose of study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition not related to the treatment of MG, including human immunodeficiency virus (HIV) infection, or a family history of congenital or hereditary immunodeficiency.
* History or evidence of administration of immunoglobulins and/or any blood products within 3 months prior to the first dose of study vaccine or a planned administration of immunoglobulins during the first 3 months of the trial.
* History or evidence of rituximab treatment within 6 months prior to first dose of study vaccine.
* History or evidence of plasmapheresis within 3 months prior to the first dose of study vaccine or a planned plasmapheresis during the first 3 months of the trial.
* At high risk for aspiration.
* Pulmonary: forced vital capacity reduced to less than 70% of predicted capacity.
* History of severe allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History or evidence of Lambert-Eaton myasthenic syndrome, drug-induced myasthenia gravis, hereditary forms of myasthenic syndrome.
* History of relevant chronic degenerative, psychiatric, or neurological disorder other than MG.
* Severe hepatic, renal or cardiac insufficiency.
* Major congenital defects or serious chronic illness other than MG.
* Positive pregnancy test or desire to become pregnant during the study.
* Female patients of child-bearing potential that do not use a reliable and highly effective method of contraception at least one month before first injection, during the study and until 3 months after the last injection.
* Any significant out-of-range Clinical Laboratory results considered as clinically significant according to Investigator's judgment.
* Previous completion or withdrawal from this study.
* Sponsor employees or investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Any medical condition that, in the opinion of the Investigator, might interfere with the subject's participation in the study, poses any added risk for the subject, or confounds the assessment of the subjects.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Safety | End of study part A (38 weeks)
  Safety assessed by laboratory tests, vital signs, electrocardiogram (ECG), adverse events, assessment of local tolerance, physical exams
Immunogenicity | End of study part A (38 weeks)
  To assess the immunogenic response after subcutaneous injections of CV-MG01 on the plasma levels of anti-peptide antibodies.

SECONDARY OUTCOMES:
Biomarker | End of study part A (38 weeks)
  To assess the effect of CV-MG01 subcutaneous injections on the plasma level of acetylcholine receptor antibodies.
Clinical efficacy | End of study part A (38 weeks)
  Clinical efficacy assessed by Quantitative MG testing Procedure extended with MG Composite Scale and MG-ADL (myasthenia gravis activities of daily living)

OTHER OUTCOMES:
Immune response | End of study part A (38 weeks)
  To explore changes in the humoral and cellular immune responses.

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Mercelis, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital, Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weathington NM, Blalock JE. Rational design of peptide vaccines for autoimmune disease: harnessing molecular recognition to fix a broken network. Expert Rev Vaccines. 2003 Feb;2(1):61-73. doi: 10.1586/14760584.2.1.61. PMID 12901598
- [Background] Galin FS, Chrisman CL, Cook JR Jr, Xu L, Jackson PL, Noerager BD, Weathington NM, Blalock JE. Possible therapeutic vaccines for canine myasthenia gravis: implications for the human disease and associated fatigue. Brain Behav Immun. 2007 Mar;21(3):323-31. doi: 10.1016/j.bbi.2006.10.001. Epub 2006 Nov 20. PMID 17113748
- See also: CuraVac: Therapeutic Vaccines for Autoimmune Diseases — http://www.curavac.com